CLINICAL TRIAL: NCT00904891
Title: Effectiveness Trial of an Adolescent Depression Prevention Program
Brief Title: Testing the Effectiveness of Adolescent Depression Prevention Programs (The OregonBlues Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH080853 (NIH); R01MH080853 (NIH); DSIR 84-CTP
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Depression
Keywords: Adolescents; Prevention; Bibliotherapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive a cognitive-behavioral group intervention.
  Interventions: Behavioral: Cognitive-behavioral group
- 2 (Active Comparator): Participants will receive cognitive-behavioral bibliotherapy.
  Interventions: Behavioral: Cognitive-behavioral bibliotherapy
- 3 (No Intervention): Participants will only complete study assessments.

INTERVENTIONS:
Behavioral: Cognitive-behavioral group — Six sessions of cognitive-behavioral depression prevention group intervention
  Arms: 1
Behavioral: Cognitive-behavioral bibliotherapy — Cognitive-behavioral bibliotherapy, delivered from the book "Feeling Good"
  Arms: 2

SUMMARY:
This study will test the effectiveness of two programs for preventing depression in adolescents.

DETAILED DESCRIPTION:
Major depression is one of the most common psychiatric disorders experienced by adolescents. Even adolescents with depressive symptoms below the level of diagnosis are at increased risk of a range of future problems, such as psychiatric disorders, impaired social functioning, and substance abuse.

Depression prevention therapies have had mixed results. Those that are implemented universally have shown little efficacy, although those that specifically target adolescents at risk of depression have shown greater efficacy. A large scale effectiveness trial-one that applies treatments outside of a lab in "real world" settings-of a targeted depression prevention therapy has not been conducted. This study will test the effectiveness of two therapies for preventing depression in adolescents. The first is a brief, group cognitive-behavioral depression prevention program, and the second is bibliotherapy, which involves giving participants a self-help book for depression. Bibliotherapy has shown efficacy in previous research but has not been examined in an effectiveness trial.

Participation in this study will last 24 months. Participants will be randomly assigned to one of three conditions: a six-session, cognitive-behavioral depression prevention group; a bibliotherapy group; and an assessment only group. Participants in the cognitive-behavioral group will meet with a study therapist and other group members to learn strategies for preventing depression. Participants in the bibliotherapy group will be given a self-help book titled "Feeling Good" with information on preventing depression. Participants in the assessment only group will receive a pamphlet on depression symptoms and treatment. All participants will complete assessments at baseline; after the cognitive-behavioral group has been completed; and at 6-, 12-, 18-, and 24-month follow-ups. These assessments will include an interview about depression symptoms and a survey about thoughts, feelings, actions, depression, and substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* High school student
* Subthreshold depressive symptoms

Exclusion Criteria:

* Meets criteria for major depression or dysthymia

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms obtained from Kiddie-Schedule for Affective Disorders and Schizophrenia (K-SADS) | Measured at baseline; post-treatment; and after 6, 12, 18, and 24 months

SECONDARY OUTCOMES:
Score on Beck Depression Inventory (BDI) | Measured at baseline; post-treatment; and after 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Rohde, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States